CLINICAL TRIAL: NCT00205582
Title: The Role of Excitatory Amino Acids on Neuronal Damage and Outcome After Traumatic Brain Injury: Assessment in Patients Using Microdialysis and (R)-[11C]PK11195 Positron Emission Tomography
Brief Title: Excitatory Amino Acids and Activated Microglia After Traumatic Brain Injury: a (R)-[11C]PK11195 PET Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001/028
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-11-04 (Estimated); Status verified 2001-05

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; PET; microglia
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Positron-Emission Tomography

INTERVENTIONS:
Device: Positron Emission Tomography

SUMMARY:
Excitatory amino acids may be involved in secondary neuronal damage after traumatic brain injury. The amount of microglia activation is an indirect measure of neuronal damage. Micorglia activation will be measured R)-[11C]PK11195 PET 1 week, 1 month and 6 months after brain injury.

DETAILED DESCRIPTION:
Glutamate and aspartate have been identified as the major excitatory neurotransmitters in the central nervous system. A massive increase in the release of these excitatory amino acids (EEA) has been described following traumatic brain injury. The resulting overstimulation of neuronal EAA receptors, particularly the N-Methyl-D-Aspartate (NMDA) receptors, leads to excessive influx of calcium through receptor gated ion-channels, causing metabolic derangement and finally cell death. Although the exact role of EEA in patients who have suffered severe head injury remains to be established, it has been shown that sustained high intracranial pressure (ICP) and poor outcome are significantly correlated to high levels of EEA using microdialysis. Disadvantages of microdialysis are that it can only be used to evaluate a limited part of the brain and that it can only be applied in the acute phase following injury. The same limits also apply to ICP measurements. Therefore, methods which evaluate both the extent and time course of damage in vivo are urgently needed.

Peripheral type benzodiazepine binding sites are a potential candidate for monitoring neuronal damage. They are not normally present in cerebral tissue, but following neuronal damage, the cells involved in the ensuing gliosis show marked expression of these sites.

(R)-PK11195 is a ligand that selectively binds to peripheral type benzodiazepine receptors. Labeled with carbon-11 its uptake can be measured with Positron Emission Tomography (PET). Thus, (R)-[11C]PK11195 PET can be used to monitor in-vivo gliosis after brain injury.

A maximum of twenty patients with traumatic brain injury will be included in this study. A microdialysis probe will be placed in the brain parenchyma to continuously measure EEA until the first PET scan is performed. Several cerebral and haemodynamic parameters, such as ICP and mean arterial blood pressure, will be registered. All patients will receive two Magnetic Resonance Imaging (MRI) scans to evaluate the extent and anatomical localization of cerebral damage. Three (R)-[11C]PK11195 PET scans will be performed: 1 week, 1 month and 6 months after the injury. Outcome will be determined using several outcome scales, including the Glasgow Outcome Scale at six months. In addition, patients will be investigated by repeated neuropsychological examinations.

ELIGIBILITY:
Inclusion Criteria:

* 1. Traumatic Brain Injury 2. Age: 18-70 years 3. Haemodynamic and respiratory stable

Exclusion Criteria:

* 1. Penetrating Skull Damage 2. Pregnancy 3. Hb < 6,5 mmol/l unless patient is known to have no history of cardiovascular disease, in which case a Hb < 5,5 mmol/l, will be the exclusion criterion 4. pH < 7,1 at initial arterial blood analysis 5. Previous neurotrauma 6. Current exposure to radiation in the workplace, or history of participation in nuclear medicine procedures, including research protocols 7. Condition which would exclude a clinical MR scan (e.g. pacemaker, shrapnel, metallic prosthesis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-05; Study Completion 2004-12

PRIMARY OUTCOMES:
Glasgow coma scale after 6 months

SECONDARY OUTCOMES:
microglia activation

CONTACTS AND LOCATIONS:
Overall Officials: Bart van Berckel, MD; PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Centre, Amsterdam, Netherlands